CLINICAL TRIAL: NCT01409798
Title: The Midwest Head and Neck Cancer Consortium Multi-Institutional Parathyroid Registry
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0324-10-EP
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Primary Hyperparathyroidism
Keywords: Hyperparathyroidism; Hypercalcemia
MeSH Terms: conditions — Hyperparathyroidism, Primary; Hyperparathyroidism; Hypercalcemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this registry is to create a database that collects clinical data to improve knowledge about primary hyperparathyroidism.

DETAILED DESCRIPTION:
This will be a multi-institutional prospective study in which patients that have undergone parathyroidectomy with intra-operative PTH assessment. The success of minimally invasive parathyroidectomy without and with intra-operative PTH will be assessed for each patient. Success for exploration without intra-operative PTH will be defined as directed exploration with detection of an abnormal parathyroid in the location suggested by imaging. Success with intra-operative PTH will be defined as per standard protocols (50% or > decrease in intra-operative PTH following excision).

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals (male and female) who have a personal diagnosis/history of primary hyperparathyroidism.
* Age 19 or greater.
* Patients who are seen and treated surgically at UNMC's Department of Otolaryngology- Head Neck Surgery .
* Able to provide informed consent.

Exclusion Criteria:

-No history of primary hyperparathyroidism

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Otolaryngology, Head and Neck Surgery clinic patients
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2010-06-09 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2015-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell B Smith, MD, Principal Investigator — University of Nebraska
Locations (6):
- United States (6):
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center, Lawrence, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - University Of Missiouri, Columbia, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sanford School of Medicine, Sioux Falls, South Dakota